CLINICAL TRIAL: NCT05378178
Title: A Phase I, Open-label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of HS-10381 in Patients With Advanced Solid Tumors
Brief Title: A PhaseⅠStudy of HS-10381 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-10381-101
Record Dates: First submitted 2022-05-06; First posted 2022-05-18 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Advanced Solid Tumor
Keywords: HS-10381; SHP2; Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase I：Dose escalation (Experimental): HS-10381 given orally QD of various dose strengths administered in 21 day dosing cycles.
  Interventions: Drug: HS-10381

INTERVENTIONS:
Drug: HS-10381 — Each subject will receive a single dose(C0) of HS-10381 and then repeat doses(C1, C2…) for 21-day cycles. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria is met.

SUMMARY:
HS-10381 is a small molecular, oral potent, SHP2 inhibitor. The first-in-human trial is conducted to assess the maximum tolerated dose (MTD) and dose limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of HS-10381 in Patients With Advanced Solid Tumors.

DETAILED DESCRIPTION:
This is a Phase 1 open-label, multicenter study to evaluate the safety, tolerability, PK and preliminary efficacy of HS-10381 in patients with advanced solid tumors by using a "3+3" dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years
2. Advanced solid tumor patients confirmed by histology or cytology for who that standard treatment is invalid, unavailable or intolerable
3. Patients have at least one target lesion according to RECEST 1.1. The requirements for target lesions are: measurable lesions without local treatment such as irradiation, or with definite progress after local treatment, with the longest diameter ≥ 10 mm in the baseline period (in case of lymph nodes, the shortest axis ≥ 15 mm is required)
4. ECOG performance status was 0-1 and did not deteriorate in the previous 2 weeks
5. Estimated life expectancy greater than (>) 12 weeks
6. Females should be using adequate contraceptive measures throughout the study; should not be breastfeeding at the time of screening, during the study and until 3 months after completion of the study; and must have evidence of non-childbearing potential
7. Sign Informed Consent Form

Exclusion Criteria:

1. Treatment with any of the following:

   1. Previous or current treatment with drugs targeting SHP2
   2. Any cytotoxic chemotherapy, investigational agents or anticancer drugs within 28 days of the first dose of study drug
   3. Radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study drug, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks of the first dose.
   4. Major surgery (including craniotomy, thoracotomy, or laparotomy, etc.) within 4 weeks of the first dose of study drug.
   5. Known and untreated, or active central nervous system metastases.
2. Existing abnormal CTCAE≥grade 2 resulted from previous treatment
3. History of other malignancy
4. Inadequate bone marrow reserve or organ function
5. Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV), unless the hepatitis is considered to be cured, Known history of HIV
6. History of hypersensitivity to any active or inactive ingredient of HS-10381.
7. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
8. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of HS-10381 | 4 weeks after initiation of treatment
  To determine the MTD of HS-10381 in subjects with advanced solid tumors.

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | Baseline through study completion(28 days after last dose)
  The CTCAE criteria will be used to assess adverse events on this trial.
Observed maximum plasma concentration (Cmax) after single dose of HS-10381 | From pre-dose to 120 hours after single dose on Cycle 0 Day 1.
  Cmax will be obtained after single dose of HS-10381 on Cycle 0 Day 1.
Observed maximum plasma concentration (Cmax ss) after multiple dose of HS-10381 | From pre-dose to 24 hours after the dose on Cycle 2 Day 1
  Cmax ss will be obtained on Cycle 2 Day 1.
Apparent terminal half-life (t1/2) after single dose of HS-10381 | From pre-dose to 120 hours after single dose on Cycle 0 Day 1
  Apparent terminal half-life is the time measured for the concentration to decrease by one half.
Area under plasma concentration versus time curve from zero to the 24-hour sampling time (AUC0-24) after single dose of HS-10381 | From pre-dose to 24 hours after single dose on Cycle 0 Day 1
  Area under the plasma concentration versus time curve from time zero to the 24-hour sampling time at which the concentration was at or above the lower limit of quantification (LLQ).
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) after single dose of HS-10381 | From pre-dose to 120 hours after single dose on Cycle 0 Day 1
  Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ).
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) after single dose of HS-10381 | From pre-dose to 120 hours after single dose on Cycle 0 Day 1
  AUC0-∞ was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the LLQ and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
To further evaluation of the anti-tumor activity of HS-10381 by assessment of objective response rate (ORR) | From the date of first occurrence of complete response (CR) or partial response (PR) on 2 consecutive occasions (≥4 weeks), until the date of disease progression or withdrawal from study，up to 2 years
  Anti-tumor efficacy will be assessed by best radiographic response based on Response Evaluation Criteria in Solid Tumors at baseline (Day -28 to -1). For patients that continue on repeating 21-Day cycles after the primary evaluation period, progression will be assessed after each 6 weeks of therapy. ORR is defined as the percentage of patients with a complete response (CR) or partial response (PR) that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Xi’an, Sichuan, China